CLINICAL TRIAL: NCT04868565
Title: Target Weaning Oxygen to Determine Duration of Caffeine for Apnea of Prematurity: a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Target Weaning Oxygen to Determine Cafffeine Duration for AOP
Acronym: DCAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wang Jianhui, Attending neonatologist, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210326
Record Dates: First submitted 2021-03-30; First posted 2021-05-03 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Apnea of Prematurity; Caffeine; Weaning Oxygen; Medicine Regimen
Keywords: apnea of prematurity; caffeine; discontinuation
MeSH Terms: conditions — Apnea | interventions — caffeine citrate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be performed by someone who are not involved in this study. Outcomes assessor will review the patients' medical record masked for the type of intervention.The investigators performing the final statistic analyses will also be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ongoing caffeine with oxygen supplement (group 1) (Experimental): samples assigned to the "ongoing caffeine with oxygen supplement (group 1)" will continue caffeine administration combining with oxygen supplement until the patients are weaned from oxygen.
  Interventions: Drug: Caffeine Citrate 20 MG/1 ML Intravenous Solution [CAFCIT]
- discontinuing caffeine with oxygen supplement (group 2) (Active Comparator): samples assigned to the "discontinuing caffeine with oxygen supplement (group 2)" will discontinue caffeine immediately after randomization, while oxygen supplement is going on.
  Interventions: Drug: Caffeine Citrate 20 MG/1 ML Intravenous Solution [CAFCIT]

INTERVENTIONS:
Drug: Caffeine Citrate 20 MG/1 ML Intravenous Solution [CAFCIT] — after randomization, caffeine citrate will be contineously prescribed to those patients assigned to the "ongoing caffeine with oxygen supplement (group 2) with a medication regimen of 10mg/kg.dose, once daily, and weekly adjustment based on the working weight.

SUMMARY:
Caffeine, a typical representative of methylxanthine, is world-widely used to manage apnea of prematurity (AOP) in neonatology. However, an appropriate medication regimen of caffeine has not been well defined until now. For example, in terms of the duration of caffeine, AAP guideline for AOP (2016) and British NICE guideline for neonatal respiratory care (2019) all recommended discontinuing caffeine when the infants reached a postmenstrual age (PMA) ≥33weeks and had a stable respiratory status, commonly manifested by weaning from non-invasive ventilation and free of apneic episodes for at least five consecutive days. Interestingly, the actual clinical settings seem to be not strictly following this recommendation. A survey of the neonatologist in North America revealed that a substantial variability existed among sites in the timing of caffeine discontinuation before discharge and the respiratory support at the time of caffeine discontinuation [1]. Another survey in Saudi Arabia also had a similar finding [2]. The optimal timing of discontinuing caffeine is still a conundrum in the field of neonatology.

Ideally, the optimal timing of discontinuing caffeine should be individual-specific. Published work has indicated that AOP and intermittent hypoxemia (IH) were frequently observed beyond 36 weeks' PMA in all gestational age groups, particularly in the 24- to 27-week infants [3, 4]. In the clinical settings, intermittent hypoxic and AOP episodes is a predominant cause of oxygen supplement in premature infants and commonly prolong the hospital stay. Optimizing arterial saturation by oxygen supplement is essential to achieve a stable cardiorespiratory status because hypoxemia could induce hypoxic sensitivity of the carotid bodies in neonates, resulting in more pronounced ventilatory depression and more frequent apneic episodes. Some RCTs have shown that continuing caffeine administration beyond PMA 34 weeks could reduce the frequency of IH episodes in premature infants [4, 5]. Therefore, theoretically, a prolonged caffeine administration over the usual duration could shorten the duration of oxygen supplements in those infants at high risk of frequent late AOP or IH. Target weaning oxygen could be an opportunistic indicator of discontinuing caffeine.

In light of the above considerations, a multicenter, retrospective, partially blinded, controlled trials will be conducted to verify the hypothesis that a novel caffeine regimen that weaning oxygen as the indicator of discontinuing caffeine could improve respiratory outcomes of very premature infants.

ELIGIBILITY:
Inclusion Criteria:

* premature infants with gestational age <30 weeks
* postmenstral age ≥32weeks
* a history of caffeine therapy
* no current positive pressure respiratory support, and free of apnea for at least five consecutive days, but still oxygen dependent
* parents or legal guardians sign informed consent to attend this study

Exclusion Criteria:

* congenital cardiorespiratory malformation, or chromosomal abnormalities
* Grade III/IV intraventricular hemorrhage, or probable brain injury attributable to confirmed central nervous system infection, severe periventricular leukomalacia or other entities;
* underwent tracheostomy
* currently on sedatives, opioids, or other medication related to depressed breath

Ages: 14 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
recurrence of apnea of prematurity (RAP) | from date of randomization until the date of discharge, assessed up to 100 days of life
  Either of the following condition is defined as a RAP event: 1. heart rate <100 beats/min; 2. weak respiratory effort requiring mask-bag ventilation; 3. A high-flow nasal cannula (HFNC) and various noninvasive and invasive ventilation are dictated by the clinical condition, where HFNC is defined as the oxygen flow is ≥2L/min; 4. Restarted caffeine therapy is considered at the discretion of the healthcare team.
duration of oxygen supplement after randomization | from date of randomization until the date of discharge, assessed up to 100 days of life
  duration of oxygen supplement after randomization
duration of hospital stay after randomization | from date of randomization until the date of discharge, assessed up to 100 days of life
  duration of hospital stay after randomization

SECONDARY OUTCOMES:
postmenstrual age of discharging home | from date of randomization until the date of discharge, assessed up to 100 days of life
  postmenstrual age at which the infants are discharged home
onset of bronchopulmonary dysplasia | from date of randomization until the date of discharge, assessed up to 100 days of life
  onset of bronchopulmonary dysplasia, defined by oxygen dependence at the postmenstrual age of 36 weeks.
severity of bronchopulmonary dysplasia | from date of randomization until the date of discharge, assessed up to 100 days of life
  evaluate the severity of bronchopulmonary dysplasia according to the 2016 NICHD proposed revision
restart caffine therapy | from date of randomization until the date of discharge, assessed up to 100 days of life
  either of the following condition considers restarting caffeine therapy: 1. RAP event requires additional interventions to positioning, suction, and tactile stimulation; 2. intermittent hypoxemia ≥ 5 episodes per day where intermittent hypoxemia is referred to as a transient desaturation with Saturation <90%, but without bradycardia; 3. restart caffeine therapy at the discretion of the healthcare team.
restart noninvasive ventilation | from date of randomization until the date of discharge, assessed up to 100 days of life
  either of the following conditions considers restarting non-invasive ventilation: 1.patients exhibit severe respiratory distress, including but not limited to tachypnea, chest indrawing, and grunting; 2. In the setting of nasal cannula oxygen supplemental, PaO2<50mmHg or SpO2<90% at the effective FiO2≥30%； 3. In the setting of incubator oxygen or hood oxygen supplement, PaO2<50mmHg or SpO2<90% at effective FiO2≥30% at the measured FiO2≥30%；4. Restart non-invasive ventilation at the discretion of the healthcare team.
reintubating the patients | from date of randomization until the date of discharge, assessed up to 100 days of life
  Either of the following conditions considers reintubating the patients: 1. Severe respiratory acidosis with PaCO2>65 mmHg and pH<7.2; 2. Refractory hypoxemia at maximal setting in the non-invasive ventilation ( SpO2< 90%, with FiO2=0.4，and PEEP reaching eight cmH2O in CPAP/NIPPV，or Paw reaching 16 cmH2O in NHFOV; 3. Severe pulmonary hemorrhage; 4. Frequent apneic episodes (≥3 episodes per hour), or at least one episode within the last 24hours requiring mask-bag ventilation, which does not respond well to methylxanthine; 5. Hemodynamic instability after a recent occurrence of neonatal resuscitation; 6. Reintubating the patients at the discretion of the healthcare team.
hospitalization cost after randomization | from date of randomization until the date of discharge, assessed up to 100 days of life
  hospitalization cost after randomization, which includes medicine cost (caffeine, and other medicine, respectively), and other healthcare cost

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, Study Director — Children's Hospital of Chongqing Medical University
Locations (41):
- China (41):
  - The First Affiliated Hospital of USTC（University of Science and Technology of China）, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Yuan Shi, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Army Military Medical University, Chongqing, Chongqing Municipality
  - Fuling Central Hospital of Chongqing City, Fuling, Chongqing Municipality
  - The People's Hospital of Dazu, Longgang, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Wanzhou, Chongqing Municipality
  - Chongqing Wanzhou Health Center for Women And Children, Wanzhou, Chongqing Municipality
  - Fuzhou Children's Hospital of Fujian Medical University, Fuzhou, Fujian
  - Xiamen Children's Hospital, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Dongguan City Maternal&Child Health Hospital, Dongguan, Guangdong
  - Maternal and Child Health Hospital of Yunfu, Yunfu, Guangdong
  - Affiliated Hospital Of Guangdong Medical University, Zhanjiang, Guangdong
  - BOAI hospital of Zhongshan, Zhongshan, Guangdong
  - Haikou Hospital of the Maternal and Child Health, Haikou, Hainan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Children's Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Hengyang Maternity and Child care hospital, Hengyang, Hunan
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - First Affiliation Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first bethune hospital of Jilin university, Changchun, Jilin
  - Qilu Children's Hospital of ShanDong University, Jinan, Shandong
  - Women & Children's Health Care Hospital of Linyi, Linyi, Shandong
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Guangyuan central hospital, Guangyuan, Sichuan
  - People's Hospital Of Leshan, Leshan, Sichuan
  - Hospital T. C. M Affiliated to Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Panzhihua Central Hospital, Panzhihua, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Kunming Children's Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Qujing City Maternal and Child Health Hospital, Qujing, Yunnan
  - The People's Hosiptal of Wenshan Prefecture, Wenshan, Yunnan
  - The First People's Hospital of Zhaotong, Zhaotong, Yunnan
  - Ningbo Women & Children's Hospital, Ningbo, Zhejiang